CLINICAL TRIAL: NCT04526938
Title: Clinical Outcomes, Radiation Dosage, and Quality of Life in Patients Treated With Fenestrated Stent Grafts for Complex Thoracoabdominal and Abdominal Aortic Aneurysms, Thoracoabdominal Aortic Aneurysms Secondary to Aortic Dissections
Brief Title: Physician-modified Endovascular Graft for Repair of Complex Thoracoabdominal and Abdominal Aortic Aneurysms
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FEVAR
Record Dates: First submitted 2020-08-21; First posted 2020-08-26 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-01

CONDITIONS: Juxtarenal Aortic Aneurysm; Suprarenal Aortic Aneurysm; Thoracoabdominal Aortic Aneurysm
Keywords: Complex Aortic Aneurysm; Complex Abdominal Aortic Aneurysm; Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal; Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Endovascular repair (Experimental): Endovascular repair of complex aortic aneurysms and thoracoabdominal aortic aneurysms including those secondary to aortic dissection using a physician-modified endovascular graft.
  Interventions: Device: Physician-Modified Cook Zenith Alpha Thoracic Endovascular Graft

INTERVENTIONS:
Device: Physician-Modified Cook Zenith Alpha Thoracic Endovascular Graft — Cook Zenith® Alpha Thoracic Endovascular Graft will be modified to allow for the maintenance of blood flow into the visceral and renal branch vessels.

SUMMARY:
The primary objective of this study is to assess the use of a physician-modified Cook Alpha Thoracic Endovascular Graft in the repair of complex aortic aneurysms and thoracoabdominal aortic aneurysms and aneurysms secondary to aortic dissections in high-risk patients having appropriate anatomy. The primary intent of the study is to assess the safety and preliminary effectiveness of the device. Additionally, the study will assess renal function, radiation exposure, and quality of life.

DETAILED DESCRIPTION:
This study is a prospective, single-center, non-randomized, single-arm study. Each enrolled subject will undergo periodic follow-up evaluations involving physical exams, computed tomography angiography (CTA) of chest, abdomen and pelvis, abdominal duplex ultrasound, creatinine measurement, quality of life questionnaire at specific, protocol-defined intervals for a period of five years following the physician-modified Cook Zenith® Alpha Endovascular Graft implant.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Life expectancy > 2 year(s)
3. Patient is considered to be at high risk of morbidity and mortality with open surgical repair
4. A patient may be entered into the study if the patient has at least one of the following:

   * Juxtarenal, suprarenal or a thoracoabdominal aortic aneurysm with a diameter ≥ 5.5 cm or 2 times the normal aortic diameter
   * Aneurysm with a history of growth ≥ 0.5 cm per year
   * Saccular aneurysms deemed at significant risk for rupture based upon physician interpretation
   * Symptomatic juxtarenal, suprarenal or a thoracoabdominal aortic aneurysm
   * Thoracoabdominal aortic aneurysms secondary to aortic dissection meeting above criteria
5. Patient is considered to be at high risk of morbidity and mortality with open surgical repair
6. Iliac or femoral access vessel morphology that is compatible with vascular access techniques, devices or accessories, with or without use of a surgical conduit
7. Nonaneurysmal aortic segment proximal to the aneurysm (neck) with a:

   * Minimum neck length of 20mm
   * Diameter in the range of 21-38mm
   * Angle less than 60° relative to the axis of the aneurysm
   * Angle less than 60° relative to the axis of the suprarenal aorta
8. Minimum branch vessel diameter greater than 5 mm
9. Iliac artery distal fixation site greater than 10mm in length and diameter in the range of 8-21mm.

Exclusion Criteria:

1. Under the age of 18 years
2. Can be treated in accordance with the instructions for use with a legally marketed endovascular prosthesis
3. Is eligible for enrollment in a manufacturer-sponsored IDE at the investigational site
4. Willing to participate in a sponsor-investigator IDE with access to a non-physician modified endovascular prostheses at the investigational site
5. Willing to travel to an investigational site with access to a non-physician modified endovascular prosthesis
6. Unwilling or unable to comply with the follow-up schedule
7. Inability or refusal to give informed consent by patient or legal representative
8. Patient is pregnant or breastfeeding
9. Life expectancy < 2-years despite successful aneurysm exclusion
10. Free rupture with hemodynamic instability
11. Ongoing infection
12. Diagnosis of, or suspected connective tissue disease
13. Known sensitivities or allergies to the materials of construction of the devices
14. Known hypersensitivity or contraindication to anticoagulation or contrast media that cannot be adequately medically managed
15. Uncorrectable coagulopathy
16. Body habitus that would inhibit x-ray visualization of the aorta or exceeds the safe capacity of the equipment
17. Patient has had a major surgical or interventional procedure unrelated to the treatment of the aneurysm planned ≤ 30 days of the endovascular repair
18. Unstable angina (defined as angina with a progressive increase in symptoms, new onset at rest or nocturnal angina)
19. Systemic or local infection that may increase the risk of endovascular graft infection
20. Leaking or free rupture of aneurysm associated with hemodynamic instability.
21. Baseline creatinine greater than 3.0 mg/dL
22. Known history of, or suspected connective tissue disorders (e.g., Marfan Syndrome, Ehler's Danlos Syndrome)

Anatomical exclusion criteria:

1. Inadequate femoral or iliac access compatible with the required delivery systems, not amenable to open surgical or endovascular conduit placement
2. Absence of a non-aneurysmal aortic segment for proximal seal zone with:

   * A diameter measured outer wall to outer wall of no greater than 38mm and no less than 21 mm;
   * Parallel aortic wall with <20% diameter change and without significant calcification and/or thrombus in the selected area of seal zone
3. Visceral vessel anatomy not compatible with physician-modified Zenith® Alpha Endovascular Graft due to excessive occlusive disease or small size not amenable to stent graft placement
4. Unsuitable distal iliac artery fixation site and anatomy:

   * Common iliac artery fixation site diameter measured outer wall to outer wall on a sectional image (CT) <8.0 mm with inability to perform open surgical conduit
   * Iliac artery diameter measured outer wall to outer wall on a sectional image (CT) >21 mm at distal fixation site, with inability to perform open internal iliac artery revascularization or iliac branch stent graft
   * Iliac artery distal fixation site <10 mm in length
   * Inability to preserve at least one hypogastric artery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Freedom from Major Adverse Events (MAE) at 30 days | 30 days
  Major Adverse Events include: Death, Bowel Ischemia, myocardial infarction, paraplegia/paraparesis, renal failure, respiratory failure, and stroke
Proportion of study subjects with treatment success at 1 year | 1 year
  Treatment success is defined as a composite of technical success and freedom from the following:
  * Aneurysm enlargement [i.e., >5mm) as compared to a preoperative CT measure using orthogonal (i.e, perpendicular to the centerline) measurements]
  * Aneurysm rupture
  * Aneurysm-related mortality
  * Conversion to open repair
  * Secondary intervention for migration, Type I and III endoleaks, device integrity failure (e.g., fracture), and patency-related events (i.e., device component stenosis or occlusion and embolic events)
Technical success | 1 year
  Technical success is defined as:
  * Successful delivery (i.e., ability to deliver the implant to the intended implantation site, without the need for unanticipated corrective intervention related to delivery) and deployment of the device at the intended location,
  * Patency of all endovascular graft and branch stent components
  * Absence of device deformations requiring unplanned placement of an additional device
  * Absence of inadvertent covering of aortic branch vessels
  * Successful withdrawal (i.e., successful withdrawal of the delivery system, without need for unanticipated corrective intervention related to withdrawal)

SECONDARY OUTCOMES:
Quality of Life measures | 30 days, 6 months; 1, 2, 3, 4 and 5 years
  Questionnaire using SF - 36™ Health Survey

CONTACTS AND LOCATIONS:
Overall Officials: Javairiah Fatima, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States